CLINICAL TRIAL: NCT00319410
Title: A New Approach to Office Hysteroscopy Compared With Traditional Hysteroscopy
Brief Title: Comparison of Two Hysteroscopy Approaches
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EWMCgyn-1
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2006-11-28 (Estimated); Status verified 2006-04

CONDITIONS: Menorrhagia
Keywords: Menorrhagia; intrauterine diagnosis; visual analogue scale
MeSH Terms: conditions — Menorrhagia

INTERVENTIONS:
Procedure: vaginoscopic hysteroscopy

SUMMARY:
This randomized clinical trial compares two methods of diagnostic hysteroscopy: vaginoscopic hysteroscopy vs. traditional method. Pain intensity was estimated using a visual analogue scale (VAS), and patient satisfaction was evaluated. These endpoints were compared by treatment assignment. Vaginoscopic hysteroscopy was associated with significantly lower VAS scores, indicating reduced experience of pain in this treatment group; however, this was not associated with improved patient satisfaction.

DETAILED DESCRIPTION:
OBJECTIVE: To compare the vaginoscopic approach of diagnostic hysteroscopy without anesthesia with the traditional diagnostic hysteroscopy after intracervical injection of Mepivacaine Hydrochloride 3%.

METHODS: A total of 130 women undergoing diagnostic hysteroscopy were included in the study and were randomized, using a computer-generated randomization list, into two groups with a ratio of 2:1. Eighty three women underwent vaginoscopy without speculum, tenaculum or anesthesia. Forty seven women received intracervical anesthesia with 10 ml of 3% mepivacaine hydrochloride solution injected at two sites (3:00 and 9:00 positions) and underwent traditional hysteroscopy using a speculum and tenaculum. Hysteroscopy was performed using a rigid 3.7 mm hysteroscope in a medium of 0.9% saline, and the image was transmitted to a screen visible to the patient. A Visual Scale Analogue (VAS) consisting of a 10 cm line was used to assess the intensity of pain experienced during and after the procedure. Overall patient satisfaction was assessed during, immediately after, 15 minutes later, and three days post hysteroscopy.

RESULTS: The mean pain score was significantly lower in the vaginoscopy group (3.8±2.7 vs 5.34±3.23, p=0.01). Patient satisfaction rate was similar in both groups.

CONCLUSION: Patients reported significantly less pain with the vaginoscopic approach to diagnostic hysteroscopy even without anesthesia compared to patients undergoing the traditional procedure with anesthesia. This new approach should therefore be considered as a replacement for the traditional hysteroscopic technique.

ELIGIBILITY:
Inclusion Criteria:adult female, referred for outpatient diagnostic hysteroscopy, subscriber to Maccabe health maintenance organization -

Exclusion Criteria:heavy vaginal bleeding; severe cervical stenosis; patients refusing the examination on an outpatient basis.

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130
Dates: Start 2005-07; Study Completion 2005-12

PRIMARY OUTCOMES:
Visual analogue scale for pain
Patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Ron Sagiv, M.D., Principal Investigator — E. Wolfson Medical Center
Locations (1):
- Maccabe Health Maintenance Organization, Tel Aviv, Israel

REFERENCES:
- [Result] Sagiv R, Sadan O, Boaz M, Dishi M, Schechter E, Golan A. A new approach to office hysteroscopy compared with traditional hysteroscopy: a randomized controlled trial. Obstet Gynecol. 2006 Aug;108(2):387-92. doi: 10.1097/01.AOG.0000227750.93984.06. PMID 16880310